CLINICAL TRIAL: NCT04370106
Title: The Impact of Frequenting a Social Leg Program on Therapeutic Adherence and Venous Leg Ulcer Wound Healing Outcomes: a Randomized Controlled Trial
Brief Title: The Impact of Frequenting a Social Leg Program on Therapeutic Adherence and Venous Leg Ulcer Wound Healing Outcomes
Acronym: legclub
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: School of Health Sciences Geneva (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: social leg program
Record Dates: First submitted 2020-04-28; First posted 2020-04-30 (Actual); Last update posted 2023-01-27 (Actual); Status verified 2023-01

CONDITIONS: Venous Leg Ulcer; Social Interaction
Keywords: leg club; education; recurrence
MeSH Terms: conditions — Varicose Ulcer; Recurrence

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Usual care for participants with existing VLU in the CG is defined as visiting the outpatient wound clinic/visits by the community care nurse as prescribed by the physician. Wound healing measurement, therapeutic adherence measurement, wound recurrence measurement, and questionnaires will be provided by the institute's nurses.
- Social leg Program (Other): Usual care as described for the CG will also be provided to the IG. Wound healing measurement, therapeutic adherence measurement, wound recurrence measurement, and questionnaires will be provided by the institute's nurses. After baseline data collection (T0) and random allocation to the intervention group, this usual care will be enhanced by frequenting a social leg program.
  Interventions: Other: Social leg program

INTERVENTIONS:
Other: Social leg program — Usual care as described for the CG will also be provided to the IG. Wound healing measurement, therapeutic adherence measurement, wound recurrence measurement, and questionnaires will be provided by the institute's nurses. After baseline data collection (T0) and random allocation to the intervention group, this usual care will be enhanced by frequenting a social leg program.
  Arms: Social leg Program

SUMMARY:
Background and rationale: Venous leg ulcers (VLU) are slow healing wounds with a recurrence rate up to 70% and a 60% risk of becoming chronic. Currently the Swiss health care system does not take in consideration social and educational needs and support for VLU patients who transition from acute care (hospital care, outpatient care) to home based self-care. To fill this gap, this study proposes to create the Social Legs Program (SLP).

Overall objectives: The objectives of the proposed study are to evaluate the impact of a frequented SLP for patients with VLU in terms of their therapeutic adherence and wound healing outcomes (wound size and wound recurrence).

Methodology of the planned study: A randomized controlled trial with 268 participants in three Swiss French institutions is proposed.

Expected results and impact: The findings of this study will generate new knowledge about support and care management of persons with VLU who transition between acute care settings and home care settings. The findings will contribute to the evidence base of clinical practice guidelines for the care of patients with VLU.

DETAILED DESCRIPTION:
Background and rationale: Venous leg ulcers (VLU) are slow healing wounds with a recurrence rate up to 70% and a 60% risk of becoming chronic. Signs and symptoms such as pain or exudate are not only a burden on those affected but also on the health care system and society in general. The estimated VLU prevalence in the general population is 3%. Treatment cost for VLU is estimated to be 4% of overall health expenditure. Current therapeutic approaches are multifaceted, focus on reducing wound size as well as preventing ulcer recurrence. Depending on the severity of the VLU treatment/care occurs in the hospital setting, outpatient setting or community setting. Currently the Swiss health care system does not take in consideration social and educational needs and support for VLU patients who transition from acute care (hospital care, outpatient care) to home based self-care. To fill this gap, this study proposes to create the Social Legs Program (SLP). This program is based on the existing Leg Club (LC) community model in the United Kingdom (UK) and will be adapted for the Swiss context. The SLP is designed to provide an environment for social interaction, peer and nursing/professional support, information sharing and personal involvement. Participation in the SLP will address the need for social and educational support in this patient group and will improve therapeutic adherence and result in enhanced wound healing as well as a reduction of the wound recurrence rate.

Overall objectives: The objectives of the proposed study are to evaluate the impact of a frequented SLP for patients with VLU in terms of their therapeutic adherence and wound healing outcomes (wound size and wound recurrence).

Specific aims: The impact of the intervention will be measured in terms of therapeutic adherence and wound healing outcomes as well as multidimensional complexity, wound assessment, patient satisfaction, depression, general nutrition, mobility and quality of sleep.

In addition, the incidence of complications (re-hospitalizations) will be measured (frequency and cost).

Methodology of the planned study: A randomized controlled trial with 268 participants in three Swiss French institutions is proposed. The study participants will be consecutive patients of the participating clinics who fulfill the inclusion criteria. Wound care will be performed according to the institutions standard clinical practice guidelines. Allocation to the intervention group (IG) or the control group (CG) will be concealed. The intervention will consist in participating in the SLP. The social program will provide patients with an opportunity to exchange and learn about the prevention measures such as the use of compression bandages, and how to prevent recurrences, and enhance healing outcomes. A study nurse, who will not be identical to the nurse in charge of the control group, will supervise this group. Due to the intervention being a social program, the study cannot be blinded for either the participants or the staff performing the intervention. The sample size assumptions are based on an adjusted (Bonferroni) two-sided alpha level of 0.05, power of 0.8, and clinically relevant effect sizes and a loss to follow up of 20%. Univariate and bivariate analysis will be conducted according to the data level.

Expected results and impact: The findings of this study will generate new knowledge about support and care management of persons with VLU who transition between acute care settings and home care settings. The findings will contribute to the evidence base of clinical practice guidelines for the care of patients with VLU. Additionally, it is in alignment with the National Strategy on the Prevention of Non-Communicable Diseases 2017 - 2024 establishing prevention work for people with enhanced risks and chronic conditions reinforcing a better social integration.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older,
* with an existing diagnosed open VLU,
* an ulcer surface <2 cm2 or having a healed VLU,
* proficiency in the French language

Exclusion Criteria:

- Valid informed consent is not or cannot be given

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 268 (Estimated)
Dates: Start 2023-12-01 (Estimated); Primary Completion 2025-03-30 (Estimated); Study Completion 2025-08-31 (Estimated)

PRIMARY OUTCOMES:
Adherence to therapy | six months
  Adherence to therapy, including physical activity, leg elevation, ankle exercises, wearing compression stockings, will be measured in minutes
Wound healing | six months
  Measurement of the impact of a social leg program on the relative reduction (in percent) of wound size in patients with VLU. Wound size will be measured using WoundWorks® imaging device
Wound recurrence | six months
  Measurement of the impact of a social leg program on absolute number of participants experiencing a recurrence (in percent) within six months over number of participants who had a healed VLU.

SECONDARY OUTCOMES:
Wound Assessment | six months
  Wound will be evaluated in terms of exudative status, smell, infection status and pain felt. The TIME strategy (T = tissue removal; I = infection control; M = moisture balance; E = edge advancement) proposed by the European Wound Management Association will be applied
Self care | six months
  Self-care score will be evaluated using the validated self care questionnaire (Venous Leg Ulcer Self-Efficacy Tool); values: minimum (0) and maximum (300); higher scores mean a better outcome.
Depression | six months
  Depression score will be evaluated using the validated geriatric depression scale questionnaire; values: minimum (0 ) and maximum (15); lower scores mean a better outcome.
Multidimensional complexity | six months
  Multidimensional complexity will be evaluated using the validated questionnaire (multidimensional complexity assessment tool, COMID): values: minimum (0 ) and maximum (30); higher scores mean a better outcome.
General nutritional status | six months
  General nutritional status of patients will be measured using the MNA® questionnaire, a validated assessment tool that identifies people malnourished or at risk of malnutrition; values: minimum ( 0) and maximum (14); higher scores mean a better outcome.
Patient Satisfaction | six months
  Patient satisfaction will be measured using the validated Patient Benefit Index (PBI) questionnaire; values: minimum (0 ) and maximum (4); higher scores mean a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Sebastian E Probst, Prof Dr, Principal Investigator — HES-SO University of Applied Sciences and Arts Western Switzerland
Locations (2):
- Switzerland (2):
  - IMAD, Carouge, Canton of Geneva
  - Cité Génération Maison de santé, Onex, Canton of Geneva

IPD SHARING:
Plan to Share IPD: No